CLINICAL TRIAL: NCT01778231
Title: Investigation of the Genetic and Environmental Determinants of MP Including Response to Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Ruth Hogg, Dr Ruth Hogg, Queen's University, Belfast
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 11/05v1
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Healthy
Keywords: Focus; uptake; Lutein; Zeaxanthin; individuals

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin Supplement (Experimental): 1 capsule of Nutrof Total made by Laboratories Thea for 16 weeks
  Interventions: Dietary Supplement: Nutrof Total
- Inert oil capsule (Placebo Comparator): 1 capsule daily for 16 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nutrof Total — Antioxidant and trace element supplement
  Arms: Vitamin Supplement
Dietary Supplement: Placebo
  Arms: Inert oil capsule

SUMMARY:
This study aims to investigate genetic and environmental determinants of macular pigment (MP) and assess the effects of lutein and zeaxanthin-rich supplements on macular pigment levels.

DETAILED DESCRIPTION:
Age-related macular degeneration is the leading cause of blindness in elderly people in western countries1. It is a degenerative condition of the macula characterized by the death or dysfunction of photoreceptors, leading to the progressive loss of central vision1. Central vision is needed for activities requiring fine vision such as reading, driving or recognizing faces. With the aging population and increasing expectations in health care it is therefore of utmost importance to preserve the quality of life and independence of the elderly through prevention of this ocular disease.

Much interest surrounds macular pigment due to its putative role in protecting the macula from oxidative stress and age-related degenerative change2, yet much is still unknown about factors that determine its uptake and deposition. Large inter-individual differences in MP have been demonstrated with several large population based studies showing that peak macular pigment density can vary by over a factor of 10 between individuals3-4. Subsequent studies have suggested a number of parameters such as age, diet, percentage body fat, gender and tobacco use5-9 as determinants of MP, however these only account for approximately a third of the variance leaving a significant proportion unexplained.

Lutein and Zeaxanthin (L and Z), constituents of MP, cannot be synthesized by the body and so are entirely dietary in origin. They are present in foods such as collard greens, spinach and Brussels sprouts10. Variation in the bitter-taste receptor gene, TAS2R38 confers the ability to taste 6-n-propylthiouracil (PROP) and phenylthiocarbamide (PTC) which is present in many of these foods11. People who taste PTC with a greater intensity are more likely to avoid these foods and therefore we hypothesize they may have lower levels of macular pigment. Thus, this study may help to identify a group at higher risk of macular degeneration.

Despite MP's dietary origin only modest correlations exist with serum and dietary levels of L and Z, and although the level of MP can be augmented in most people by diet or supplementation the response is variable and not always correlated with baseline level. Most supplementation studies identify a sub-group of "retinal non-responders"12 in which serum values of the carotenoids have risen, yet no change is found in macular pigment, the reason for this is not clear. The first part of our study will provide a well-phenotyped group in which to explore this further. Several studies have also shown that peak macular pigment levels are strongly heritable13-14 suggesting genetics may play an important role. Although no gene has currently been clearly identified the ApoE gene has been suggested to show an association with macular pigment level. A supplementation study in this population will be able to determine whether the genes identified on a cross-sectional basis do determine uptake of the nutritional supplement. We may also be able to identify specific demographic or lifestyle factors of non-responders which may help to explain the phenomenon.

1. Carpentier S, Knaus M, Suh M. Associations between Lutein, Zeaxanthin, and Age-Related Macular Degeneration: An Overview. Clinical Reviews in Food Science and Nutrition. 2009 49:313-326
2. Whitehead AJ, Mares J, Danis RP. Macular Pigment: A Review of Current Knowledge. Arch Opthamol. July 2006; 124: 1038-1045
3. Ciulla TA, Curran-Celantano J, Cooper DA, et al. Macular pigment optical density in a midwestern sample. Ophthalmology. Apr 2001;108(4):730-737.
4. Hammond BR, Jr., Caruso-Avery M. Macular pigment optical density in a Southwestern sample. Invest Ophthalmol Vis Sci. May 2000;41(6):1492-1497.
5. Hammond BR, Jr., Curran-Celentano J, Judd S, et al. Sex differences in macular pigment optical density: relation to plasma carotenoid concentrations and dietary patterns. Vision Res. Jul 1996;36(13):2001-2012.
6. Hammond BR, Jr., Wooten BR, Snodderly DM. Cigarette smoking and retinal carotenoids: implications for age-related macular degeneration. Vision Res. Sep 1996;36(18):3003-3009.
7. Ciulla TA, Hammond BR, Jr. Macular pigment density and aging, assessed in the normal elderly and those with cataracts and age-related macular degeneration. Am J Ophthalmol. Oct 2004;138(4):582-587.
8. Curran-Celentano J, Hammond BR, Jr., Ciulla TA, Cooper DA, Pratt LM, Danis RB. Relation between dietary intake, serum concentrations, and retinal concentrations of lutein and zeaxanthin in adults in a Midwest population. Am J Clin Nutr. Dec 2001;74(6):796-802.
9. Nolan J, O'Donovan O, Kavanagh H, et al. Macular pigment and percentage of body fat. Invest Ophthalmol Vis Sci. Nov 2004;45(11):3940-3950.
10. Carpentier S, Knaus M, Suh M. Associations between Lutein, Zeaxanthin, and Age-Related Macular Degeneration: An Overview. Critical Reviews in Food Science and Nutrition. 2009; 49(4): 313-326
11. Bachmanov A, Beauchamp G. Taste Receptor Genes. Annual Review of Nutrition. 2007.27:389-414
12. Hammond BR, Jr., Johnson EJ, Russell RM, et al. Dietary modification of human macular pigment density. Invest Ophthalmol Vis Sci. Aug 1997;38(9):1795-1801.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers,
* male or female,
* aged 18-50 years

Exclusion Criteria:

* evidence of eye disease,
* inability to give informed written consent,
* any other health problem which would interfere with ability to adhere to the study protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Macular Pigment Measurement | 16 weeks
  Macular Pigment Measurement using Heterochromatic Flicker Photometry

SECONDARY OUTCOMES:
Serum Lutein and Zeaxanthin | 16 weeks
Macular Pigment (reflectometry) | 16 weeks
  Macular Pigment level measured using reflectometry

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Public Health, Belfast, Antrim, United Kingdom